CLINICAL TRIAL: NCT03737708
Title: Compare Efficacy and Safety Between Biologics + Methotrexate (MTX) vs Biologics + Tacrolimus (TAC) (Switched From Biologics + Methotrexate (MTX)) in the Patients With Rheumatoid Arthritis (RA): Randomized, Interventional, Open, Active Controlled, Parallel Group, Multicenter-designed, Phase 4 Clinical Trial
Brief Title: A Study Comparing Biologics + Methotrexate With Biologics + Tacrolimus in Patients With Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 506-MA-3187
Record Dates: First submitted 2018-11-08; First posted 2018-11-09 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: tacrolimus; abatacept; Prograf; adalimumab; methotrexate; tocilizumab; FK506
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Tacrolimus; Methotrexate; Adalimumab; tocilizumab; Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tacrolimus + biologics (Experimental): Participants will receive tacrolimus daily for 12 weeks. In addition, each participant will be administered one of adalimumab, tocilizumab, or abatacept for 12 weeks.
  Interventions: Drug: tacrolimus; Biological: adalimumab; Biological: tocilizumab; Biological: abatacept
- methotrexate + biologics (Active Comparator): Participants will receive methotrexate weekly for 12 weeks. In addition, each participant will be administered one of adalimumab, tocilizumab, or abatacept for 12 weeks.
  Interventions: Drug: methotrexate; Biological: adalimumab; Biological: tocilizumab; Biological: abatacept

INTERVENTIONS:
Drug: tacrolimus — Administered orally
  Other Names: FK506; Prograf
  Arms: tacrolimus + biologics
Drug: methotrexate — Administered orally
  Arms: methotrexate + biologics
Biological: adalimumab — Administered as subcutaneous injection
Biological: tocilizumab — Administered by intravenous injection
Biological: abatacept — Administered by intravenous injection

SUMMARY:
The purpose of this study is to compare the efficacy of Biologics + Methotrexate with Biologics + Tacrolimus measured by the disease activity score 28 (DAS28) erythrocyte sedimentation rate (ESR) and the American College of Rheumatology (ACR) scores. The study will also assess the safety of the combinations.

DETAILED DESCRIPTION:
This study will include 4-weeks screening and a 12-week open-label treatment period.The participants in this study will visit the center five (5) times over the study period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with rheumatoid arthritis (RA) diagnosed by the 2010 American College of Rheumatology/European League Against Rheumatism (ACR/EULAR).
* Subjects who have been treated with combination therapy of one of biologic agent (adalimumab, tocilizumab, or abatacept) + methotrexate (MTX) over 2 months prior to Visit 1.
* Disease Activity Score (DAS28) erythrocyte sedimentation rate (ESR) ≥ 3.2 at screening and baseline.
* Subject agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Subjects with a past history of allergic reaction to Investigational Product or Comparative Drug used in this study.
* Subjects who were given tacrolimus (TAC) within three months before participation in this study.
* Subjects who have been treated with combination therapy of one of biologic agent (adalimumab, tocilizumab, or abatacept) + MTX exceeds 3 months at Baseline.
* Subjects who were already taking 20 mg of MTX at Screening Period.
* Subjects who were given the prohibited concomitant medications prior to randomization.
* Subjects with a medical history of clinically significant blood, gastrointestinal, endocrine, lung, nerve, or brain diseases at screening.
* Subjects with a medical history of clinically significant liver, kidney, or heart diseases:

  * Liver disease: Aspartate Aminotransferase (AST) and Alanine aminotransferase (ALT) > 3 × upper limit of normal (ULN) at screening, viral infection, nonviral infection, and liver cirrhosis;
  * Kidney disease: serum creatinine > 2.0 mg/dL at screening;
  * Heart disease: heart failure of ≥ The New York Heart Association class 3, arrhythmia or ischemic heart disease requiring treatment, and QTc interval > 450 ms on Electrocardiogram (ECG) at screening;
* Subjects with a history of uncontrolled diabetes (glycosylated hemoglobin > 8.5%).
* Subjects with hyperkalemia or serum potassium level > ULN of site reference ranges at screening.
* Subjects with severe respiratory disease or chronic generalized infectious disease.
* Subject who have a history of chronic infection or severe or life-threatening infection within 24 weeks before the baseline visit.
* Subject who are known to be infected by Human Immunodeficiency Virus, Hepatitis B, or Hepatitis C.
* Subject has a history of active tuberculosis or latent tuberculosis infection without treatment.
* Subject with mental disorder uncontrolled by drugs.
* Subject with chronic diarrhea, ulcerative stomatitis, gastric ulcer, or ulcerative colitis.
* Subject with genetic disorders including galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.
* Subject with maculopathy, retinal disorders, or clinically significant eye diseases that may lead to visual disorder.
* Subject with bone marrow disorder, leukopenia, and blood cell disorder such as severe anemia and thrombocytopenia.
* Subject with a history of major surgery within 12-weeks before screening.
* Subject who were diagnosed with malignant tumors within 5 years before screening or who need treatment for malignant tumors diagnosed in the past.
* Patients with basal cell and squamous cell carcinomas of the skin or carcinoma in situ of the cervix uteri that has been excised and cured, may be included on the study at the discretion of the investigator.
* Female subject who is positive for the serum pregnancy test at Visit 1 among a woman of childbearing potential (WOCBP) (menopausal is defined as amenorrhea for at least one year) or not surgically sterile, or is not willing to use appropriate contraception during the study. Female subject trying to become pregnant or is currently pregnant or breast feeding.
* Male subject who donates sperm during the treatment period and for at least 30 days whichever is longer after the final study drug administration.
* Male subject with a pregnant or breastfeeding partner(s) who do not agree to remain abstinent or use a condom for the duration of the pregnancy, or for the time partner is breastfeeding, throughout the study period and for 30 days whichever is longer after the final study drug administration.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-06-16 (Actual); Study Completion 2020-06-16 (Actual)

PRIMARY OUTCOMES:
Change in disease activity score 28 (DAS28) erythrocyte sedimentation rate score (ESR) score at 12 weeks | From baseline (week 1) to week 12
  DAS28-ESR will be calculated using data from tender joint count (TJC) (28 joints), swollen joint count (SJC) (28 joints), ESR and Subject's Global Assessment of Arthritis (SGA) with the formula; DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 x SGA.
  High disease activity: DAS28 score exceeding 5.1 Moderate disease activity: DAS28 score of exceeding 3.2 to 5.1 Low disease activity: DAS28 score of less than or equal to 3.2 If the DAS28 score is less than 2.6, the participant will be considered to be in DAS28 remission.

SECONDARY OUTCOMES:
Disease activity score 28 (DAS28) erythrocyte sedimentation rate (ESR) rate score at 4 weeks | At 4 weeks
  DAS28-ESR will be calculated using data from TJC (28 joints), SJC (28 joints), ESR and SGA with the formula; DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 x SGA.
  High disease activity: DAS28 score exceeding 5.1 Moderate disease activity: DAS28 score of exceeding 3.2 to 5.1 Low disease activity: DAS28 score of less than or equal to 3.2 If the DAS28 score is less than 2.6, the participant will be considered to be in DAS28 remission.
DAS28 (ESR) score at 8 weeks | At 8 weeks
  DAS28-ESR will be calculated using data from TJC (28 joints), SJC (28 joints), ESR and SGA with the formula; DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 x SGA.
  High disease activity: DAS28 score exceeding 5.1 Moderate disease activity: DAS28 score of exceeding 3.2 to 5.1 Low disease activity: DAS28 score of less than or equal to 3.2 If the DAS28 score is less than 2.6, the participant will be considered to be in DAS28 remission.
DAS28 (ESR) score at 12 weeks | At 12 weeks
  DAS28-ESR will be calculated using data from TJC (28 joints), SJC (28 joints), ESR and SGA with the formula; DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 x SGA.
  High disease activity: DAS28 score exceeding 5.1 Moderate disease activity: DAS28 score of exceeding 3.2 to 5.1 Low disease activity: DAS28 score of less than or equal to 3.2 If the DAS28 score is less than 2.6, the participant will be considered to be in DAS28 remission.
Change in DAS28 (ESR) score at 4 weeks | From baseline (week 1) to week 4
  DAS28-ESR will be calculated using data from TJC (28 joints), SJC (28 joints), ESR and SGA with the formula; DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 x SGA.
  High disease activity: DAS28 score exceeding 5.1 Moderate disease activity: DAS28 score of exceeding 3.2 to 5.1 Low disease activity: DAS28 score of less than or equal to 3.2 If the DAS28 score is less than 2.6, the participant will be considered to be in DAS28 remission.
Change in DAS28 (ESR) score at 8 weeks | From baseline (week 1) to week 8
  DAS28-ESR will be calculated using data from TJC (28 joints), SJC (28 joints), ESR and SGA with the formula; DAS28- ESR = 0.56√(TJC) + 0.28√(SJC) + 0.70 ln ESR + 0.014 x SGA.
  High disease activity: DAS28 score exceeding 5.1 Moderate disease activity: DAS28 score of exceeding 3.2 to 5.1 Low disease activity: DAS28 score of less than or equal to 3.2 If the DAS28 score is less than 2.6, the participant will be considered to be in DAS28 remission.
ACR 20 response rate | At 12 weeks
  Percent of participants with American College of Rheumatology (ACR) 20 response rate The ACR20 response requires that all criteria from (1) to (3) be met compared with Week 0 (baseline); (1), Tender Joint Count (TJC) >= 20% reduction; (2), Swollen Joint Count (SJC) >= 20% reduction;(3) >= 20% improvement in three or more of the following five parameters - [1] subject's assessment of pain, [2] Subject's Global Assessment of Arthritis (SGA), [3] Physician's Global Assessment of Arthritis (PGA), [4] health assessment questionnaire-disability index (HAQ-DI), [5] acute phase reactant (erythrocyte sedimentation rate (ESR)).
ACR50 response rate | At 12 weeks
  Percent of participants with ACR50 response rate The ACR50 response indicates a 50% improvement in all criteria used in the ACR20 assessment.
ACR70 response rate | At 12 weeks
  Percent of participants with ACR70 response rate The ACR70 response indicates a 70% improvement in all criteria used in the ACR70 assessment.
Safety assessed by Adverse Events (AEs) | Up to 16 weeks
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product.
Safety assessed by incidence of serious adverse events (SAE) | Up to 16 weeks
  Adverse Event (AE) is considered "serious" if the investigator or sponsor view any of the following outcomes: Death, life-threatening, persistent or significant disability/incapacity, congenital anomaly or birth defect, hospitalization, or medically important event.
Safety assessed by incidence of treatment emergent adverse events (TEAE) | Up to 12 weeks
  Treatment Emergent Adverse Event (TEAE) is defined as any AE which starts, or worsens, after the first dose of study drug through 30 days after the last dose of study drug.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) | Up to 16 weeks
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and /or adverse events (AEs) | Up to 16 weeks
  Number of participants with potentially clinically significant vital sign values.
Number of participants with physical exam abnormalities and/or adverse events (AEs) | Up to 16 weeks
  Number of participants with potentially clinically significant physical exam values.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Korea, Inc.
Locations (10):
- South Korea (10):
  - Site KR82003, Daegu
  - Site KR82007, Daegu
  - Site KR82006, Daejeon
  - Site KR82002, Incheon
  - Site KR82009, Seongnam
  - Site KR82001, Seoul
  - Site KR82005, Seoul
  - Site KR82010, Seoul
  - Site KR82012, Seoul
  - Site KR82013, Suwon

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/patientStudySearch.aspx?RID=;;;506-MA-3187